CLINICAL TRIAL: NCT02412722
Title: A Phase 1, Open-label Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MLN0128 (an Oral mTORC 1/2 Inhibitor) as a Single Agent and in Combination With Paclitaxel in Adult Patients With Advanced Nonhematologic Malignancies
Brief Title: A Safety, Tolerability, and Pharmacokinetics Study of MLN0128 as a Single Agent and in Combination With Paclitaxel in Adults With Advanced Nonhematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MLN0128-1004; U1111-1161-4803 (Registry Identifier: WHO)
Record Dates: First submitted 2015-03-10; First posted 2015-04-09 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Non-hematologic Malignancy
Keywords: Drug therapy
MeSH Terms: interventions — sapanisertib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Single-Agent QD Arm: Sapanisertib 3 mg (Experimental): Following Pharmacokinetic (PK) - Run in Period, sapanisertib 3 mg milled capsules, orally, once, daily in a 28-day Cycle, under fasted conditions, starting from Cycle 2 for up to 9 cycles. The dose of sapanisertib was modified based on safety and tolerability during each 28-day cycle.
  Interventions: Drug: Sapanisertib
- Single-Agent QD Arm: Sapanisertib 4 mg (Experimental): Following PK Run-In Period, sapanisertib 4 mg milled capsules, orally, once, daily in a 28-day Cycle, under fasted conditions, for up to 13 cycles.
  Interventions: Drug: Sapanisertib
- Combination Arm: Sapanisertib 4 mg + Paclitaxel 80 mg/m^2 (Experimental): Sapanisertib 4 mg milled capsules, orally, once, for 3 consecutive days following each paclitaxel administration (Days 2-4, 9-11, 16-18, and 23-25) in a 28-day Cycle, under fasted conditions, for up to 12 cycles, and paclitaxel 80 mg/m^2, intravenously (IV), on Days 1, 8, and 15 in 28-day Cycle, for up to 6 cycles.
  Interventions: Drug: Sapanisertib; Drug: Paclitaxel
- Combination Arm: Sapanisertib 6 mg + Paclitaxel 80 mg/m^2 (Experimental): Sapanisertib 6 mg milled capsules, orally, once, for 3 consecutive days following each paclitaxel administration (Days 2-4, 9-11, 16-18, and 23-25) in a 28-day Cycle, under fasted conditions, for up to 9 cycles, and paclitaxel 80 mg/m^2, IV, on Days 1, 8, and 15 in 28-day Cycle, for up to 9 cycles. The dose of sapanisertib was modified based on safety and tolerability during each 28-day cycle.
  Interventions: Drug: Sapanisertib; Drug: Paclitaxel
- Single-Agent QW Arm: Sapanisertib 20 mg (Experimental): Sapanisertib 20 mg, capsules milled API, QW in a 28-day Cycle, for up to 6 cycles.
  Interventions: Drug: Sapanisertib
- Single-Agent QW Arm: Sapanisertib 30 mg (Experimental): Sapanisertib 30 mg, capsules, milled API, QW in a 28-day Cycle, for up to 10 cycles.
  Interventions: Drug: Sapanisertib

INTERVENTIONS:
Drug: Sapanisertib — Sapanisertib capsules
Drug: Paclitaxel — Paclitaxel injection
  Arms: Combination Arm: Sapanisertib 4 mg + Paclitaxel 80 mg/m^2; Combination Arm: Sapanisertib 6 mg + Paclitaxel 80 mg/m^2

SUMMARY:
The purposes of this study are to evaluate the safety and tolerability of sapanisertib (MLN0128) milled active pharmaceutical ingredient (API) capsules administered both as a single agent and in combination with paclitaxel, to characterize the effect of a high-fat meal on the pharmacokinetics (PK) of sapanisertib milled API capsules, and to characterize the PK of sapanisertib milled API capsules when administered on an empty stomach approximately 24 hours after paclitaxel infusion.

DETAILED DESCRIPTION:
The drug being tested in this study is called sapanisertib (MLN0128). Sapanisertib is being tested to assess its safety and tolerability when administered alone or in combination with paclitaxel in people who have nonhematologic malignancies. Sapanisertib is also being tested to characterize its PK properties (how is processed by the body) when administered with a high-fat meal compared to on an empty stomach. This study will look at side effects and lab results in people who take sapanisertib with or without paclitaxel.

This open label study enrolled 61 patients. Participants receiving only sapanisertib will participate in a 6-day PK Run-In Period where sapanisertib 4 mg capsules are administered under fasted conditions on Days 1 and 4, and with a high-fat breakfast on Day 3. The main treatment period will begin within 14 days from Day 6 of the PK Run-In Period. In the main treatment period participants will receive sapanisertib 4 mg daily in a 28-day Cycle for up to 12 cycles. Participants in the treatment arm receiving sapanisertib and paclitaxel will not have a PK Run-In Period and will receive sapanisertib 6 mg daily on Days 2-4, 9-11, 16-18, and 23-25 in a 28-day Cycle for up to 12 cycles and paclitaxel 80 mg/m^2 intravenously (IV) on Days 1, 8, and 15 in 28-day Cycle, for up to 12 cycles. The dose of sapanisertib may be modified based on safety and tolerability during each 28-day cycle in either treatment arm.

This multi-centre trial will be conducted in the United States. The overall time to participate in this study is up to 15 months. Participants in the sapanisertib only arm will make up to 32 visits to the clinic and participants in the sapanisertib and paclitaxel arm will make up to 26 visits to the clinic. All participants will make a final visit to the clinic 30 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age is ≥ 18 years, including males and females.
2. Has Advanced nonhematologic malignancies, with the exception of primary brain tumor, and have failed or are not eligible for standard of care therapy. History of brain metastasis may be allowed if all the following criteria are met: brain metastases have been treated, there is no evidence of progression or hemorrhage after treatment, dexamethasone discontinued for ≥ 4 weeks before first study drug administration, and there is no ongoing requirement for dexamethasone or anti-epileptic drugs.
3. Has received not more than 4 prior lines of systemic cytotoxic chemotherapy for advanced or metastatic disease.
4. Has Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 1.
5. Has adequate organ function, including the following:

   * Bone marrow reserve consistent with absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L; platelet count ≥ 100 x 10^9/L; and hemoglobin ≥ 9 g/dL without transfusion in the last 2 weeks
   * Hepatic: total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN), transaminases (aspartate aminotransferase [AST]/serum glutamic oxaloacetic transaminase [SGOT] and alanine aminotransferase [ALT]/serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases are present)
   * Renal: normal serum creatinine or calculated creatinine clearance ≥ 60 mL/min based either on Cockcroft-Gault estimate or based on urine collection (12- or 24-hour)
   * Metabolic: fasting serum glucose (≤ 130 mg/dL) and fasting triglycerides ≤ 300 mg/dL
6. Has left ventricular ejection fraction (LVEF) within 5 absolute percentage points of institutional standard of normal as measured by echocardiogram (ECHO) or multiple gated acquisition scan (MUGA) within 4 weeks before first study drug administration (ie, if the institutional normal is 50%, participant's LVEF may be as low as 45% to be eligible for the study).
7. Is a female participants who:

   * Are postmenopausal for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, or
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)

   Male participants, even if surgically sterilized (ie, status postvasectomy), who:
   * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, or
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods for the female partner] and withdrawal are not acceptable methods of contraception.)
8. Has ability to swallow oral medications.
9. Has voluntary written consent obtained before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.

Exclusion Criteria:

1. Has a diagnosis of primary brain tumor.
2. Has untreated brain metastasis or history of leptomeningeal disease or spinal cord compression.
3. Has failed to recover from the reversible effects of prior anticancer therapies with the exception of alopecia, and after-effects associated with prior tyrosine kinase inhibitor therapy, such as hair depigmentation, hypothyroidism, and/or splinter hemorrhage.
4. Has received prior cancer therapy or other investigational therapy within 2 weeks before the first administration of study drug. For prior therapies with a half-life longer than 3 days, the interval must be at least 28 days before the first administration of study drug, and the participant must have documented disease progression.
5. Has initiation of hematopoietic growth factors within 1 week before the first administration of any study drug; participants already receiving hematopoietic growth factors on a chronic basis for ≥ 4 weeks are eligible.
6. Has chronic systemic corticosteroid (except inhalers) use within 1 week before the first administration of study drug. Premedication with dexamethasone before paclitaxel administration in this study is allowed.
7. Has manifestations of malabsorption due to prior gastrointestinal surgery, gastrointestinal disease, or for an unknown reason that may alter the absorption of MLN0128.
8. Has poorly controlled diabetes mellitus defined as glycosylated hemoglobin (HbA1c) > 7%; participants with a history of transient glucose intolerance due to corticosteroid administration are allowed if all other eligibility criteria are met.
9. Has other clinically significant comorbidities, such as uncontrolled pulmonary disease, active central nervous system disease, active infection, or any other condition that could compromise the participant's participation in the study.
10. Has a known human immunodeficiency virus infection.
11. Is pregnant (positive serum or urine pregnancy test) or breastfeeding.
12. Has any history of unstable angina, myocardial infarction, New York Heart Association Class III or IV heart failure, and/or pulmonary hypertension.
13. Has significant active cardiovascular disease including:

    * Uncontrolled high blood pressure (ie, systolic blood pressure > 180 mmHg, diastolic blood pressure > 95 mmHg)
    * Grade 3 or higher valvular disease
    * Grade 3 or higher atrial fibrillation
    * Grade 3 or higher bradycardia
    * Endocarditis
    * Pulmonary embolism
    * Recent cerebrovascular accident/transient ischemic attack ≤ 6 months before enrollment
14. Diagnosed or treated for another malignancy within 2 years before the first dose or previously diagnosed with another malignancy and have any evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
15. Single-Agent QD Arm participants participating in the pharmacokinetic (PK) Run-In (only): participants who use proton pump inhibitors (PPIs) less than 5 days before the first MLN0128 PK Run-In dose OR use H2 receptor antagonists within 24 hours of the first PK Run-In dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-03-26 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (5):
- United States (5):
  - Scottsdale, Arizona
  - Sarasota, Florida
  - Oklahoma City, Oklahoma
  - Germantown, Tennessee
  - Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Background] Chopra M. Annual Congress of the European Society for Medical Oncology (ESMO): Copenhagen, Denmark; 7-11 October 2016. Target Oncol. 2016 Dec;11(6):705-709. doi: 10.1007/s11523-016-0464-3. No abstract available. PMID 27812901
- [Derived] Moore KN, Bauer TM, Falchook GS, Chowdhury S, Patel C, Neuwirth R, Enke A, Zohren F, Patel MR. Phase I study of the investigational oral mTORC1/2 inhibitor sapanisertib (TAK-228): tolerability and food effects of a milled formulation in patients with advanced solid tumours. ESMO Open. 2018 Feb 1;3(2):e000291. doi: 10.1136/esmoopen-2017-000291. eCollection 2018. PMID 29464110

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in United States from 26 March 2015 to 31 May 2018.
Pre-assignment Details: Participants were enrolled in 3 cohorts in the study: 1)Single-Agent QD Arm, 2)Combination Arm and 3)Single-Agent QW Arm. Participants in Single-Agent QD Arm first completed pharmacokinetic (PK) run-in period, to assess the effect of dosing condition (ie, fed vs fasted) and manufacturing process (ie, milled vs unmilled API) on PK of sapanisertib.
Groups:
- Single-Agent QD Arm: Sapanisertib 3 mg: Following Pharmacokinetic (PK) - Run in Period, sapanisertib 3 mg milled capsules, orally, once, daily in a 28-day Cycle, under fasted conditions, starting from Cycle 2 for up to 9 cycles.
- Single-Agent QD Arm: Sapanisertib 4 mg: Following PK Run-In Period, sapanisertib 4 mg milled capsules, orally, once, daily in a 28-day Cycle, under fasted conditions, starting from Cycle 2 for up to 13 cycles.
- Combination Arm: Sapanisertib 6 mg + Paclitaxel 80 mg/m^2: Sapanisertib 6 mg milled capsules, orally, once, for 3 consecutive days following each paclitaxel administration (Days 2-4, 9-11, 16-18, and 23-25) in a 28-day Cycle, under fasted conditions, for up to 9 cycles, and paclitaxel 80 mg/m^2, IV, on Days 1, 8, and 15 in 28-day Cycle, for up to 9 cycles.
Period: Overall Study
Arm/Group | Single-Agent QD Arm: Sapanisertib 3 mg | Single-Agent QD Arm: Sapanisertib 4 mg | Combination Arm: Sapanisertib 4 mg + Paclitaxel 80 mg/m^2 | Combination Arm: Sapanisertib 6 mg + Paclitaxel 80 mg/m^2 | Single-Agent QW Arm: Sapanisertib 20 mg | Single-Agent QW Arm: Sapanisertib 30 mg
Started | 11 | 8 | 7 | 15 | 7 | 13
Safety Population | 11 | 6 | 7 | 15 | 7 | 13
Completed (Completed=Participants who completed study treatment.) | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 11 | 8 | 7 | 15 | 7 | 13
Not completed — Adverse Event | 0 | 2 | 0 | 3 | 0 | 3
Not completed — Progressive Disease | 6 | 4 | 4 | 9 | 3 | 3
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 2 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Received drug in run-in and discontinued | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Reason not Specified | 3 | 0 | 2 | 1 | 2 | 6

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Single-Agent QD Arm: Sapanisertib 3 mg | Single-Agent QD Arm: Sapanisertib 4 mg | Combination Arm: Sapanisertib 4 mg + Paclitaxel 80 mg/m^2 | Combination Arm: Sapanisertib 6 mg + Paclitaxel 80 mg/m^2 | Single-Agent QW Arm: Sapanisertib 20 mg | Single-Agent QW Arm: Sapanisertib 30 mg | Total
Number analyzed (Participants) | 11 | 8 | 7 | 15 | 7 | 13 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (15.76) | 60.5 (8.17) | 56.2 (7.75) | 63.4 (12.74) | 57.0 (16.45) | 60.5 (12.02) | 60.7 (12.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 5 | 11 | 3 | 10 | 44
  Male | 2 | 2 | 2 | 4 | 4 | 3 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 11 | 8 | 7 | 14 | 6 | 12 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 2 | 1 | 1 | 7
  White | 9 | 7 | 6 | 11 | 5 | 11 | 49
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 8 | 7 | 15 | 7 | 13 | 61
Height [Mean (Standard Deviation); unit: cm] | 163.9 (7.78) | 168.0 (8.52) | 170.2 (6.68) | 166.0 (11.43) | 165.3 (11.92) | 164.4 (5.05) | 165.9 (8.76)
Weight [Mean (Standard Deviation); unit: kg] | 71.2 (17.02) | 74.4 (14.11) | 87.2 (35.23) | 75.3 (27.45) | 63.3 (15.55) | 61.8 (11.10) | 71.6 (21.96)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug. An SAE is defined as an untoward medical occurrence, significant hazard, contraindication, side effect or precaution that at any dose: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: From Day 1, Cycle 1 through 30 days after the last dose of study drug (up to 15 months)
Population: Safety population included participants who received at least 1 dose of study drug. PK-Run In population included participants who received more than one dose of study drug in PK Run-In period.
Measure: Count of Participants; unit: Participants
Groups:
- PK-Run In Period Fasted (Unmilled): Sapanisertib, 4 mg, unmilled capsules, orally, QD under fasted conditions on Day 1 in 14-day PK Run-In Period prior to Cycle 1, Day 1.
- PK-Run In Period Fed (Milled): Sapanisertib, 4 mg, milled capsules, orally, QD, under fed conditions on Day 3 in 14-day PK Run-In Period prior to Cycle 1, Day 1.
- PK-Run In Period Fasted (Milled): Sapanisertib, 4 mg, milled capsules, orally, QD under fasted conditions on Day 5 in 14-day PK Run-In Period prior to Cycle 1, Day 1.
Arm/Group | PK-Run In Period Fasted (Unmilled) | PK-Run In Period Fed (Milled) | PK-Run In Period Fasted (Milled) | Single-Agent QD Arm: Sapanisertib 3 mg | Single-Agent QD Arm: Sapanisertib 4 mg | Combination Arm: Sapanisertib 4 mg + Paclitaxel 80 mg/m^2 | Combination Arm: Sapanisertib 6 mg + Paclitaxel 80 mg/m^2 | Single-Agent QW Arm: Sapanisertib 20 mg | Single-Agent QW Arm: Sapanisertib 30 mg
Number analyzed (Participants) | 19 | 19 | 17 | 11 | 6 | 7 | 15 | 7 | 13
Participants
  At least one AE | 7 | 6 | 9 | 11 | 6 | 7 | 14 | 6 | 13
  Serious AE | 1 | 0 | 2 | 3 | 2 | 2 | 7 | 4 | 7

2. Primary Outcome: Geometric Mean Ratio of Cmax: Maximum Observed Plasma Concentration of Sapanisertib Milled Active Pharmaceutical Ingredient (API) Capsules Under Fasted and Fed Conditions
Time Frame: Days 3 and 5 predose and at multiple time points (up to 24 hours) post-dose
Population: PK population included participants with protocol specified dosing and conditions and PK data to reliably estimate PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Sapanisertib 4 mg Milled Capsules Under Fed Conditions: Sapanisertib 4 mg milled capsules, orally, once, after a high-fat breakfast, on Days 3 and 5.
- Sapanisertib 4 mg Milled Capsules Under Fasted Conditions: Sapanisertib 4 mg unmilled capsules, orally, once, under fasted conditions, on Days 3 and 5.
Arm/Group | Sapanisertib 4 mg Milled Capsules Under Fed Conditions | Sapanisertib 4 mg Milled Capsules Under Fasted Conditions
Number analyzed (Participants) | 19 | 17
ng/mL | 21.6 (37.4) | 36.4 (50.6)
Statistical Analysis 1: Comparison: Sapanisertib 4 mg Milled Capsules Under Fed Conditions vs Sapanisertib 4 mg Milled Capsules Under Fasted Conditions; Test type: Superiority; Geometric Mean Ratio = 0.59, 90% CI 2-sided [0.46 to 0.76]

3. Primary Outcome: Geometric Mean Ratio of AUC(0-last): Area Under the Plasma Concentration Curve From Time Zero to the Time of the Last Quantifiable Concentration of Sapanisertib Milled API Capsules Under Fasted and Fed Conditions
Time Frame: Days 3 and 5 predose and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Sapanisertib 4 mg Milled Capsules Under Fed Conditions | Sapanisertib 4 mg Milled Capsules Under Fasted Conditions
Number analyzed (Participants) | 19 | 17
ng*hr/mL | 205.9 (59.8) | 229.2 (58.2)
Statistical Analysis 1: Comparison: Sapanisertib 4 mg Milled Capsules Under Fed Conditions vs Sapanisertib 4 mg Milled Capsules Under Fasted Conditions; Test type: Superiority; Geometric Mean Ratio = 0.90, 90% CI 2-sided [0.59 to 1.36]

4. Primary Outcome: Geometric Mean Ratio of AUC(0-inf): Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity for Sapanisertib Milled API Capsules Under Fasted and Fed Conditions
Time Frame: Days 3 and 5 predose and at multiple time points (up to 24 hours) post-dose
Population: PK population included participants with protocol specified dosing and conditions and PK data to reliably estimate PK parameters. Overall number of participants analyzed is the number of participants with the data available for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Sapanisertib 4 mg Milled Capsules Under Fed Conditions | Sapanisertib 4 mg Milled Capsules Under Fasted Conditions
Number analyzed (Participants) | 13 | 13
ng*hr/mL | 382.8 (64.7) | 369.2 (50.0)
Statistical Analysis 1: Comparison: Sapanisertib 4 mg Milled Capsules Under Fed Conditions vs Sapanisertib 4 mg Milled Capsules Under Fasted Conditions; Test type: Superiority; Geometric Mean Ratio = 1.04, 90% CI 2-sided [0.72 to 1.49]

5. Primary Outcome: Cmax: Maximum Observed Plasma Concentration of Sapanisertib Milled API Capsules Under Fasted Conditions Approximately 24 Hours After Paclitaxel Infusion
Time Frame: Cycle 1, Day 2 pre-dose and at multiple time points (up to 8 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Combination Arm: Sapanisertib 4 mg + Paclitaxel 80 mg/m^2 | Combination Arm: Sapanisertib 6 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 7 | 15
ng/mL | 35.2 (22.33) | 71.4 (29.16)

6. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration of Sapanisertib Milled API Capsules Under Fasted Conditions Approximately 24 Hours After Paclitaxel Infusion
Time Frame: Cycle 1, Day 2 pre-dose and at multiple time points (up to 8 hours) post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Combination Arm: Sapanisertib 4 mg + Paclitaxel 80 mg/m^2 | Combination Arm: Sapanisertib 6 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 7 | 15
hours | 2.2 [0.9 to 5.6] | 1.1 [0.5 to 3.0]

7. Primary Outcome: AUC(0-8): Area Under the Plasma Concentration Curve From Time Zero to 8 Hours Post-dose for Sapanisertib Milled API Capsules Under Fasted Conditions Approximately 24 Hours After Paclitaxel Infusion
Time Frame: Cycle 1, Day 2 pre-dose and at multiple time points (up to 8 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Combination Arm: Sapanisertib 4 mg + Paclitaxel 80 mg/m^2 | Combination Arm: Sapanisertib 6 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 7 | 15
ng*hr/mL | 144.8 (84.15) | 260.6 (89.59)

8. Secondary Outcome: Geometric Mean Ratio of Cmax: Maximum Observed Plasma Concentration of Sapanisertib Milled Versus Unmilled API Capsules Under Fasted Conditions
Time Frame: Days 1 and 3 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Sapanisertib 4 mg Milled Capsules Under Fasted Conditions: Sapanisertib 4 mg Milled capsules, orally, once, under fasted conditions, on Days 1 and 3.
- Sapanisertib 4 mg Unmilled Capsules Under Fasted Conditions: Sapanisertib 4 mg unmilled capsules, orally, once, under fasted conditions, on Days 1 and 3.
Arm/Group | Sapanisertib 4 mg Milled Capsules Under Fasted Conditions | Sapanisertib 4 mg Unmilled Capsules Under Fasted Conditions | Single-Agent QW Arm: Sapanisertib 20 mg | Single-Agent QW Arm: Sapanisertib 30 mg
Number analyzed (Participants) | 17 | 19 | 7 | 13
ng/mL | 36.4 (50.6) | 34.0 (48.1) | 208.6 (17.3) | 235.2 (43.4)
Statistical Analysis 1: Comparison: Sapanisertib 4 mg Milled Capsules Under Fasted Conditions vs Sapanisertib 4 mg Unmilled Capsules Under Fasted Conditions; Test type: Superiority; Geometric Mean Ratio = 1.07, 90% CI 2-sided [0.78 to 1.47]

9. Secondary Outcome: Geometric Mean Ratio of AUC(0-last): Area Under the Plasma Concentration Curve From Time Zero to the Time of the Last Quantifiable Concentration for Sapanisertib Milled Versus Unmilled API Capsules Under Fasted Conditions
Time Frame: Days 1 and 3 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Sapanisertib 4 mg Milled Capsules Under Fasted Conditions | Sapanisertib 4 mg Unmilled Capsules Under Fasted Conditions | Single-Agent QW Arm: Sapanisertib 20 mg | Single-Agent QW Arm: Sapanisertib 30 mg
Number analyzed (Participants) | 17 | 19 | 7 | 13
hr*ng/mL | 229.2 (58.2) | 204.6 (57.3) | 1238.1 (53.3) | 1528.8 (43.5)
Statistical Analysis 1: Comparison: Sapanisertib 4 mg Milled Capsules Under Fasted Conditions vs Sapanisertib 4 mg Unmilled Capsules Under Fasted Conditions; Test type: Superiority; Geometric Mean Ratio = 1.12, 90% CI 2-sided [0.75 to 1.68]

10. Secondary Outcome: AUC(0-inf): Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity for Sapanisertib Milled Versus Unmilled API Capsules Under Fasted Conditions
Time Frame: Days 1 and 3 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Sapanisertib 4 mg Milled Capsules Under Fasted Conditions | Sapanisertib 4 mg Unmilled Capsules Under Fasted Conditions | Single-Agent QW Arm: Sapanisertib 20 mg | Single-Agent QW Arm: Sapanisertib 30 mg
Number analyzed (Participants) | 13 | 13 | 7 | 13
hr*ng/mL | 369.2 (50.0) | 400.8 (48.2) | 1326.2 (61.5) | 1636.6 (45.2)
Statistical Analysis 1: Comparison: Sapanisertib 4 mg Milled Capsules Under Fasted Conditions vs Sapanisertib 4 mg Unmilled Capsules Under Fasted Conditions; Test type: Superiority; Geometric Mean Ratio = 0.92, 90% CI 2-sided [0.67 to 1.26]

11. Secondary Outcome: Overall Response Rate Based on Response Evaluation Criteria in Solid Tumors (RECIST)
Description: ORR is defined as the percentage of participants with complete response (CR) or partial response (PR) using Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. CR: Disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR: At least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions.
Time Frame: Baseline then every 2 cycles beginning at Cycle 3, Day 1, until disease progression, death or end of study (Up to 14 months)
Population: Safety population included participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Single-Agent QD Arm: Sapanisertib 3 mg | Single-Agent QD Arm: Sapanisertib 4 mg | Combination Arm: Sapanisertib 4 mg + Paclitaxel 80 mg/m^2 | Combination Arm: Sapanisertib 6 mg + Paclitaxel 80 mg/m^2 | Single-Agent QW Arm: Sapanisertib 20 mg | Single-Agent QW Arm: Sapanisertib 30 mg
Number analyzed (Participants) | 11 | 6 | 7 | 15 | 7 | 13
percentage of participants | 9.1 | 16.7 | 14.3 | 20.0 | 0.0 | 0.0

12. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of first study drug administration to the date of first documented PD or death due to any cause. PD was based on response evaluation criteria in solid tumors (RECIST V1.1), defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: as for outcome 11
Population: Data was not collected for this outcome measure.
Arm/Group | Single-Agent QD Arm: Sapanisertib 3 mg | Single-Agent QD Arm: Sapanisertib 4 mg | Combination Arm: Sapanisertib 4 mg + Paclitaxel 80 mg/m^2 | Combination Arm: Sapanisertib 6 mg + Paclitaxel 80 mg/m^2 | Single-Agent QW Arm: Sapanisertib 20 mg | Single-Agent QW Arm: Sapanisertib 30 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Clinical Benefit Response (CBR)
Description: CBR is defined as the percentage of participants with complete response (CR) or partial response (PR) or stable disease (SD) using Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. CR: Disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR: At least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions. SD is neither shrinkage by greater than or equal to 30% of the sum of the longest diameter of target lesions or the increase of lesions by greater than or equal to 20% of the sum of the longest diameter of target lesions.
Time Frame: as for outcome 11
Population: Safety population included participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Single-Agent QD Arm: Sapanisertib 3 mg | Single-Agent QD Arm: Sapanisertib 4 mg | Combination Arm: Sapanisertib 4 mg + Paclitaxel 80 mg/m^2 | Combination Arm: Sapanisertib 6 mg + Paclitaxel 80 mg/m^2 | Single-Agent QW Arm: Sapanisertib 20 mg | Single-Agent QW Arm: Sapanisertib 30 mg
Number analyzed (Participants) | 11 | 6 | 7 | 15 | 7 | 13
percentage of participants
  CR+PR+SD | 63.6 | 33.3 | 42.9 | 53.3 | 42.9 | 46.2
  CR + PR + SD (>= 6 Months) | 36.4 | 33.3 | 14.3 | 26.7 | 0.0 | 7.7

14. Secondary Outcome: Change From Baseline in Tumor Volume/Size
Description: Changes in tumor size and volume will be determined by measurements from computed tomography (CT) and magnetic resonance imaging (MRI) scans.
Time Frame: From Cycle 1 Day -14 to 14 months
Population: Data was not collected for this outcome measure.
Arm/Group | Single-Agent QD Arm: Sapanisertib 3 mg | Single-Agent QD Arm: Sapanisertib 4 mg | Combination Arm: Sapanisertib 4 mg + Paclitaxel 80 mg/m^2 | Combination Arm: Sapanisertib 6 mg + Paclitaxel 80 mg/m^2 | Single-Agent QW Arm: Sapanisertib 20 mg | Single-Agent QW Arm: Sapanisertib 30 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days post last dose (Up to 15 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. PK-Run In population included participants who received more than one dose of study drug in PK Run-In period.
Arm/Group | PK-Run In Period Fasted (Unmilled) | PK-Run In Period Fed (Milled) | PK-Run In Period Fasted (Milled) | Single-Agent QD Arm: Sapanisertib 3 mg | Single-Agent QD Arm: Sapanisertib 4 mg | Combination Arm: Sapanisertib 4 mg + Paclitaxel 80 mg/m^2 | Combination Arm: Sapanisertib 6 mg + Paclitaxel 80 mg/m^2 | Single-Agent QW Arm: Sapanisertib 20 mg | Single-Agent QW Arm: Sapanisertib 30 mg
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/17 | 0/11 | 1/6 | 0/7 | 1/15 | 0/7 | 1/13
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/19 | 2/17 | 3/11 | 2/6 | 2/7 | 7/15 | 4/7 | 7/13
Other Adverse Events (participants affected / at risk) | 7/19 | 6/19 | 9/17 | 11/11 | 6/6 | 7/7 | 14/15 | 6/7 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PK-Run In Period Fasted (Unmilled) (N=19) | PK-Run In Period Fed (Milled) (N=19) | PK-Run In Period Fasted (Milled) (N=17) | Single-Agent QD Arm: Sapanisertib 3 mg (N=11) | Single-Agent QD Arm: Sapanisertib 4 mg (N=6) | Combination Arm: Sapanisertib 4 mg + Paclitaxel 80 mg/m^2 (N=7) | Combination Arm: Sapanisertib 6 mg + Paclitaxel 80 mg/m^2 (N=15) | Single-Agent QW Arm: Sapanisertib 20 mg (N=7) | Single-Agent QW Arm: Sapanisertib 30 mg (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with sapanisertib 30 mg and is not related.
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with sapanisertib 6 mg + paclitaxel 80 mg/m^2 and is not related.
Enterococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Clostridium test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adenoid cystic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with sapanisertib 4 mg and is not related.
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PK-Run In Period Fasted (Unmilled) (N=19) | PK-Run In Period Fed (Milled) (N=19) | PK-Run In Period Fasted (Milled) (N=17) | Single-Agent QD Arm: Sapanisertib 3 mg (N=11) | Single-Agent QD Arm: Sapanisertib 4 mg (N=6) | Combination Arm: Sapanisertib 4 mg + Paclitaxel 80 mg/m^2 (N=7) | Combination Arm: Sapanisertib 6 mg + Paclitaxel 80 mg/m^2 (N=15) | Single-Agent QW Arm: Sapanisertib 20 mg (N=7) | Single-Agent QW Arm: Sapanisertib 30 mg (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eyelid irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 5 | 1 | 5 | 6 | 4 | 6
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 4 | 5 | 8 | 4 | 2
Vomiting (Gastrointestinal disorders) | 4 | 1 | 2 | 3 | 1 | 2 | 5 | 2 | 7
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 4 | 4 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 1 | 2 | 2 | 2 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 4 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 6 | 4 | 2 | 9 | 3 | 8
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site rash (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 1 | 4 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Systemic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 2 | 0 | 0 | 2 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hear rate irregular (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymph node palpable (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 4 | 2 | 3 | 8 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 2 | 1 | 3 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 3 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Balance Disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mental Impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 3 | 2 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thinking abnormal (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Micturition Urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 6 | 3 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4 | 0 | 2 | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Pain Of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retension (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Study Protocol (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/22/NCT02412722/Prot_000.pdf
  • Statistical Analysis Plan (2015-08-12): https://cdn.clinicaltrials.gov/large-docs/22/NCT02412722/SAP_001.pdf